CLINICAL TRIAL: NCT04197700
Title: PRotocolized vs pErsonalized Blood preSSUre peRi-operative paramEters in Coronary Artery Bypass Grafting Surgery: The PRESSURE CABG Cardiac Surgery Trial
Brief Title: The PRESSURE CABG Cardiac Surgery Trial
Acronym: PRESSURECABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00095074
Record Dates: First submitted 2019-12-03; First posted 2019-12-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Bypass Grafting; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Pragmatic, prospective, single-center, unit-based cluster crossover, open-label registry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Arm (Other): Personalized Arm: The target MAP will be defined as +/- 5% of the resting MAP. Resting MAP will be defined in priority order using one of the following MAP measurements:
  * Pre-operative anesthesia or surgical consultation;
  * Other physician outpatient consultation (e.g. cardiology, family physician, internist) within 30 days of surgery;
  * Inpatient measurement the night before surgery;
  * Pre-anesthetic MAP
  The order of the measurements prioritizes outpatient MAPs given that temporary pre-operative discontinuation of anti-hypertensive agents could potentially raise, while fasting and/or fluid restriction pre-operatively could potentially lower resting blood pressure.39 The lower and upper safety limits of personalized MAP targets will be 50mmHg and <90mmHg, respectively.
  Interventions: Other: Target MAP Management
- Protocolized Arm (Other): Protocolized Arm: The target MAP will be defined as 65 +/- 5mmHg. Pharmacologic and fluid treatment decisions will be at the discretion of the most responsible physician.
  In both study arms, the blood pressure control period will extend from anesthetic induction until 12 hours after admission to the CSICU. As an additional safety metric, the anesthesiologist will be encouraged to utilize clinically-driven cerebral saturation monitoring to identify potential hypoperfusion. In cases with low bilateral saturations where the anesthesiologist feels low MAP may be the putative mechanism, the investigators will request that MAPs be raised in 5mmHg increments. Following completion of the study protocol, the MAP and/or systolic blood pressure targets will be at the discretion of the most responsible physician.
  Interventions: Other: Target MAP Management

INTERVENTIONS:
Other: Target MAP Management — Target MAP Management

SUMMARY:
This study will be a pragmatic, prospective, single-centre, unit-based cluster crossover, open-label registry trial. The cardiac surgical intensive care unit (CSICU) will be cluster assigned to alternating MAP targets in 6-month blocks in a sequence. Additional sites across Alberta may be added, as necessary.

DETAILED DESCRIPTION:
Personalized Arm: The target MAP will be defined as +10% of the resting MAP. Resting MAP will be defined in priority order using one of the following MAP measurements:

* Pre-operative anesthesia or surgical consultation;
* Other physician outpatient consultation (e.g. cardiology, family physician, internist) within 30 days of surgery;
* Inpatient measurement the night before surgery;
* Pre-anesthetic MAP

The lower and upper safety limits of personalized MAP targets will be 50mmHg and <90mmHg, respectively.

Protocolized Arm: The target MAP will be defined as 65 +/- 5mmHg. Pharmacologic and fluid treatment decisions will be at the discretion of the most responsible physician.

In both study arms, the blood pressure control period will extend from anesthetic induction until 12 hours after admission to the CSICU. As an additional safety metric, the anesthesiologist will be encouraged to utilize clinically-driven cerebral saturation monitoring to identify potential hypoperfusion. In cases with low bilateral saturations where the anesthesiologist feels low MAP may be the putative mechanism, the investigators will request that MAPs be raised in 5mmHg increments. Following completion of the study protocol, the MAP and/or systolic blood pressure targets will be at the discretion of the most responsible physician.

ELIGIBILITY:
Inclusion Criteria:

* All patients > or = to 18 years of age undergoing non-emergent CABG

Exclusion Criteria:

* Pre-induction use of intravenous inotrope, vasopressor, or vasodilator
* Re-operation during the index hospital stay
* Non-CABG valvular or aortic surgery
* *Patients with end-stage renal disease or pre-operative AKI (defined as in-hospital increase in creatinine by >50%) will be excluded from the renal outcomes but included in the analysis of secondary outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Composite of delirium or AKI | within 7 days of surgery
  composite of delirium(defined as Intensive care delirium screening checklist score >=4) or Acute kidney injury (defined as a >=50% rise in serum creatinine)m
Re-operation for bleeding | Within 7 days of surgery
  re-operation for bleeding

SECONDARY OUTCOMES:
Delirium | Through 7 days
  Incidence (defined as Intensive care delirium screening checklist score >=4) and duration of Delirium (in days)
The incidence of Stroke | Up to the time of hospital discharge, estimated average 5 days
  post-operative stroke
Renal Outcomes | Up to the time of hospital discharge, estimated average 5 days
  Risk of Acute kidney injury, Acute Kidney Injury, Renal Failure, Renal replacement therapy according to RIFLE criteria
Difference in peak median creatinine levels | Up to the time of hospital discharge, estimated average 5 days
  Absolute difference in peak median creatinine levels
Chest tube output | Through 48 hours post-op
  Median differences in chest tube output
Blood Products | Through 48 hours post-operatively
  Number of red blood cell, fresh frozen plasma, and platelet transfusions
IV Vasoactive Support | Up to the time of ICU discharge, , estimated average 2 days
  Median duration of intravenous vasoactive support
Vasoactive support >24hrs | Up to 25 hours post-operatively
  Percentage of patients with vasoactive support >24 hours
Mechanical Ventilation | Up to the time of ICU discharge, estimated average 4 hours
  Duration of mechanical ventilation
Length of Stay | Up to the time of ICU discharge, estimated average 2 days
  Duration of CSICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No